CLINICAL TRIAL: NCT01092156
Title: Prenatal Breastfeeding Education to Reduce Nipple Pain
Acronym: BEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Association of American Medical Colleges (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 200614137-5; MM-0844-05/05 (Other Grant/Funding Number: American Association of Medical Colleges)
Record Dates: First submitted 2010-03-22; First posted 2010-03-24 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Nipple Pain During Lactation
Keywords: Nipple pain during lactation
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Education on Infant-led latching (Active Comparator)
  Interventions: Behavioral: Education
- Standard education (No Intervention)

INTERVENTIONS:
Behavioral: Education — Education on Infant-led latching
  Arms: Education on Infant-led latching

SUMMARY:
This study is a randomized controlled trial to evaluate the effectiveness of different approaches to prenatal teaching of infant latch.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who intend to breastfeed their infants
* Single infant
* Resides in catchment area
* Has phone
* Speaks English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Nipple pain day 3 postpartum | Day 3 postpartum

SECONDARY OUTCOMES:
Breastfeeding status day 30 postpartum | Day 30 postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Caroline J Chantry, M.D., Principal Investigator — University of California, Davis; Kathryn G Dewey, Ph.D., Principal Investigator — University of California, Davis
Locations (1):
- Sutter Davis Hospital, Davis, California, United States